CLINICAL TRIAL: NCT03648801
Title: A Post-marketing Surveillance to Assess Safety and Efficacy of Telostop Plus Tab.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-TAR-P401
Record Dates: First submitted 2018-08-14; First posted 2018-08-27 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hypertension, Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertention, Dyslipidemia: NA (Observation study)

SUMMARY:
Post-marketing surveillance of Telostop Plus Tab.

DETAILED DESCRIPTION:
This study will collect clinical data, mainly focused on safety, in Korean population as per the requirement of MFDS for market authorization.

ELIGIBILITY:
Inclusion Criteria:

* The patient who is first prescribed and administered Telostop plus Tab.

Exclusion Criteria:

* The patients who are overreacting to this drug or its components
* The patients with severe renal impairment

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patient diagnosed with hypertention and dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event after this drug administration in general medical practice | 24 weeks
  Any adverse events occurred after this drug dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.
Incidence of serious adverse event after this drug administration in general medical practice | 24 weeks
  Any serious adverse events occurred after this drug dosing will be recorded. Description of serious adverse event(s) including type of serious adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the serious adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be serious adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be serious adverse events.